CLINICAL TRIAL: NCT05210816
Title: The Effect of Acceptance and Commitment Therapy on Psychotic Symptoms and Functioning Levels in Early Psychosis Patients
Brief Title: Acceptance and Commitment Therapy (ACT) in Early Psychosis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SY200217B09
Record Dates: First submitted 2022-01-13; First posted 2022-01-27 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2022-01

CONDITIONS: Acceptance and Commitment Therapy; Psychotic Disorders; Psychiatric Nursing
Keywords: Acceptance and Commitment Therapy; Early psychosis; Psychotic symptom; Functionality; Psychiatric Nursing; Early intervention
MeSH Terms: conditions — Psychotic Disorders | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Intervention Model Description: Intervention and control group
Who Masked: Participant
Masking Description: Experimental: Intervention group ''Acceptance and Commitment Therapy Based Intervention Program was applied to the intervention group Intervention: Behavioral: Acceptance and Commitment Therapy No Intervention: Control group Only data collection was carried out. No attempt was made by the researcher during the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACT (Experimental): ''Acceptance and Commitment Therapy (ACT) Based Intervention Program was applied to the intervention group.
  Interventions: Behavioral: Acceptance and Commitment Therapy
- Control (No Intervention): Only data collection was carried out. No attempt was made by the researcher during the study.

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy — Acceptance and Commitment Therapy Based Intervention Program was applied to the intervention group in eight sessions online. Each session will last an average of 60-90 minutes. There will be two sessions for one group per week.
  Arms: ACT

SUMMARY:
This study is to examine the effect of Acceptance and Commitment Therapy applied to patients in early psychosis patients on psychotic symptoms and functionality levels.

DETAILED DESCRIPTION:
This study is a pretest, posttest, follow-up, randomized controlled experimental study. This study will be conducted at the Health Sciences University Sultan II. Abdulhamid Han Training and Research Hospital, Department of Psychiatry. According to the G-power analysis results, the minimum sample size of the study was calculated as 40 (intervention 20, control 20). Before randomization, the Personal Information Form and P1-P3 questions on the Positive and Negative Syndrome Scale (PANNS) will be applied to the patients in order to identify the patients with early psychosis. Computer-aided https://www.random.org/integers/ program will be used to assign the intervention and control group without bias. It is planned that the intervention group will consist of at least 8 participants and the program will be implemented as three intervention groups. Acceptance and Commitment Therapy (ACT) Based Intervention Program was applied to the intervention group in eight sessions online. Each session will last an average of 60-90 minutes. There will be two sessions for one group per week. The control group will not receive any intervention by the researcher, and participants will continue with their routine treatment plan. The intervention groups after the program is completed and three months later, follow-up will be done by applying the post-test, while the control group will be followed-up by applying the post-test four weeks and three months later.

In the preparation of the interventions and planning of the sessions based on ACT, the researcher utilised studies in the literature and the basic ACT training she had received. After preparation of the ACT intervention protocol, it was given its final shape by obtaining the views of specialists working in this field. The sessions were prepared based on six components of psychological flexibility found at the basis of ACT.

ELIGIBILITY:
Inclusion Criteria:

* The consent of himself/herself or his/she guardian to participate in the research,
* Being diagnosed with schizophrenia and other psychotic disorders for a minimum of six months and a maximum of three years according to DSM-V diagnostic criteria,
* Not to be in the acute attack period of the disease,
* The home environment is suitable for online conversation (computer/smartphone, internet at home, the patient can be alone in the room during the session, etc.)
* Being between the ages of 18-65,
* Ability to read and write,
* There is no communication problem at a level that prevents the conversation,
* Absence of mental retardation, neurocognitive disorder, alcohol and substance abuse

Exclusion Criteria:

* Her/his is or her/his is guardian's refusal to participate in the research,
* Being diagnosed with schizophrenia and other psychotic disorders for less than six months or for more than three years, according to DSM-V diagnostic criteria,
* Being in the acute attack period of the disease,
* Not being able to read and write,
* Having a communication problem at a level that prevents the conversation,
* Having mental retardation, neurocognitive disorder, alcohol and substance addiction

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Positive and Negative Syndrome Scale (PANSS) | 9 month
  The PANNS scale provides an assessment of the severity of psychotic symptoms. Data is collected by the researcher through a semi-structured interview with the patients. In the scale consisting of 30 spiritual parameters; seven of them belong to the positive symptoms subscale, seven to the negative symptoms subscale, and the remaining sixteen to the general psychopathology subscale. The total score varies between 30-210. A total score of 58-74 from the scale is defined as mild, 75-94 points as moderate, 95-115 points as marked disease, and 116 and above points as severe disease.

SECONDARY OUTCOMES:
Social Functioning Assessment Scale | 9 month
  It is a 19-item Likert-type scale developed for schizophrenia patients. Each item is in the range of 1-3 points. It is seen that the scale consists of four factors as interpersonal relations and entertainment, self-care, independent living skills and working life. The score that can be obtained from the scale is in the range of 19-57, and a high score from the scale means that the individual has a high level of social functionality.

CONTACTS AND LOCATIONS:
Overall Officials: Duygu ÖZER, MsN, Principal Investigator — Saglik Bilimleri Universitesi
Locations (1):
- Saglik Bilimleri Universitesi, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ozer D, Dissiz M. The effect of online group based acceptance and commitment therapy on psychotic symptoms and functioning levels of individuals with early psychosis. Schizophr Res. 2024 May;267:55-64. doi: 10.1016/j.schres.2024.03.018. Epub 2024 Mar 22. PMID 38518479